CLINICAL TRIAL: NCT00169767
Title: Holmium Laser Ablation of the Prostate (HoLAP) Versus KTP Laser Vaporization of the Prostate: A Randomized Comparison Study
Brief Title: Holmium Laser Ablation of the Prostate (HoLAP) Versus KTP Laser Vaporization of the Prostate
Status: Terminated | Type: Observational
Why Stopped: Poor enrollment
Sponsor: Indiana Kidney Stone Institute (Other)
Collaborators: Lumenis Be Ltd. (Industry)
Responsible Party: James E. Lingeman, M.D., Indiana Kidney Stone Institute
Other Study IDs: 05-042
Record Dates: First submitted 2005-09-09; First posted 2005-09-15 (Estimated); Last update posted 2008-04-25 (Estimated); Status verified 2008-04

CONDITIONS: Benign Prostatic Hyperplasia
Keywords: Enlarged Prostate; BPH
MeSH Terms: conditions — Prostatic Hyperplasia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- A: Comparison study between KTP and HoLAP procedures for BPH
  Interventions: Other: Comparison study between KTP and HoLAP for BPH

INTERVENTIONS:
Other: Comparison study between KTP and HoLAP for BPH — Comparison study between KTP and HoLAp for BPH
  Other Names: BPH

SUMMARY:
Many options currently exist to relieve the symptoms caused by benign prostatic hyperplasia (BPH). At present, transurethral resection of the prostate (TURP) serves as the surgical standard to which all other operative treatments are compared. Although TURP provides excellent short and long-term results, this procedure has many potential risks and complications. The desire to avoid the potential risks of TURP and still achieve results of comparable durability has led to the development of alternative surgical procedures.

One such surgical alternative in the treatment of BPH is holmium laser ablation of the prostate (HoLAP). HoLAP has been compared to TURP in a randomized clinical trial with comparable outcomes in both uroflow rate and symptom score improvements (Mottet, et al 1999). Use of the holmium laser in treating BPH provides specific advantages over TURP. The risk of dilutional hyponatremia is eliminated, as the holmium laser can be used in conjunction with a normal saline irrigant. In addition, the hemostatic properties of the holmium laser results in superior hemostasis, thus minimizing the risk of bleeding. HoLAP has been utilized for prostate glands up to 60 grams in volume, as larger glands become more inefficient to treat using a tissue vaporization technique.

Recently, another laser technology has been introduced for the surgical treatment of BPH, the potassium titanyl-phosphate (KTP) laser. This modality can also be used to vaporize obstructive prostate tissue, and has been studied through single arm clinical studies. Short-term results are promising, with significant improvements in voiding symptoms and urine flow rates as well as minimal associated morbidity. However, to date a randomized comparison study between HoLAP and KTP laser vaporization of the prostate has not been reported. A group of investigators with extensive experience with both procedures intends to objectively compare these two procedures in a randomized clinical trial.

DETAILED DESCRIPTION:
The traditional surgical therapy for BPH is a transurethral resection of the prostate (McConnell et al, 1994). This surgery involves the insertion of a telescope (resectoscope) transurethrally into the prostate and bladder. An electrocautery loop attached to the resectoscope is then used to core out the inside of the prostate until the surgical capsule of the prostate is reached. A large catheter is left in the bladder for at least 1 day and saline irrigation of the bladder is often required for post-operative bleeding. Once the urine is clear, the catheter is removed and the patient undergoes a voiding trial. If voiding is successful, the patient is discharged home.

TURP produces excellent short and long-term results and remains a standard of care for the surgical treatment of BPH. Unfortunately, this durable procedure has many potential risks and complications including bleeding requiring blood transfusion (~5%), intraoperative complications (e.g. prostate capsule perforation), urethral and bladder injury, dilutional hyponatremia and the TUR syndrome, urinary tract infection (~5-10%), incontinence (~1%), erectile dysfunction (~5%), bladder neck contracture or urethral stricture (~5%), and delayed bleeding resulting in clot retention or secondary procedures to control bleeding. (American Urological Association [AUA] Guideline on Management of Benign Hyperplasia (2003). Chapter 1: Diagnosis and Treatment Recommendations Journal of Urology, 170: 530, 2003.)

One alternative to TURP that has been shown in a randomized clinical trial to reproduce the excellent results of TURP has been holmium laser ablation of the prostate (HoLAP) (Mottet et al, 1999). HoLAP is a simple procedure to perform in smaller prostate glands (ideally < 60 gm) and recently reported results suggest that this procedure produces good results that are durable up to 7 years (Gilling et al, 2002).

A new technology for use during prostate ablation is the high power potassium titanyl-phosphate (KTP) laser (Malek et al, 2000). This surgical procedure involves the use of the Laserscope™ KTP laser (San Jose, CA) to vaporize obstructing prostatic tissue in a technique similar to HoLAP. Most investigators have reported no significant complications with this new technology and in most cases, significant improvements in American Urological Association symptom scores and urine flow rates have been documented (Malek et al, 2000). Unfortunately, no randomized comparison study between HoLAP and KTP laser prostatectomy has been performed.

ELIGIBILITY:
Inclusion Criteria:

* Ability to give informed consent
* Lower urinary tract symptoms (LUTS) felt to be secondary to bladder outlet obstruction from benign prostatic hyperplasia
* Maximum urinary flow rate < 15 ml/sec, voided volume ≥ 125 cc
* American Urological Association symptom score ≥ 9
* Transrectal ultrasound determined prostate volume ≤ 60 cc

Exclusion Criteria:

* Inability to give informed consent
* Maximum urinary flow rate ≥ 15 ml/sec
* Transrectal ultrasound determined prostate volume > 60cc
* AUA symptom score < 9
* Active urinary tract infection
* Bleeding diathesis
* Neurological disease that is felt to affect the bladder or a history of a neurogenic or chronically decompensated bladder
* Known prostate cancer
* Active bladder cancer (within the last 2 years)
* Prostate specific antigen (PSA) > 4.0 unless previous negative biopsy
* Urinary retention
* Post-void residual (PVR) > 300 cc

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: urology clinic
Sampling Method: Probability Sample
Enrollment: 18 (Actual)
Dates: Start 2005-05; Primary Completion 2008-04 (Actual); Study Completion 2008-04 (Actual)

PRIMARY OUTCOMES:
operative parameters, short and long-term results, and complications associated with HoLAP and KTP laser vaporization of the prostate | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: James E Lingeman, MD, Principal Investigator — Methodist Urology, LLC
Locations (3):
- United States (3):
  - Methodist Hospital, Indianapolis, Indiana
  - Oakwood Annapolis Hospital, Westland, Michigan
  - Duke University, Durham, North Carolina